CLINICAL TRIAL: NCT05038982
Title: Efficacy, Safety, and Tolerability of Abrocitinib for Reducing Pruritus in Adults With Prurigo Nodularis and Chronic Pruritus of Unknown Origin
Brief Title: Efficacy of Abrocitinib for Reducing Pruritus in Adults With Prurigo Nodularis and Chronic Pruritus of Unknown Origin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Duke University (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00262268
Record Dates: First submitted 2021-08-23; First posted 2021-09-09 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Prurigo Nodularis; Pruritus; Chronic Pruritus; Chronic Prurigo; Skin Diseases
MeSH Terms: conditions — Pruritus; Skin Diseases | interventions — abrocitinib

STUDY DESIGN:
Intervention Model Description: This is a non-randomized study with two arms conducted in parallel: an arm of 10 Prurigo Nodularis (PN) patients, and an arm of 10 Chronic pruritus of unknown origin (CPUO) patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prurigo Nodularis (Experimental): Prurigo Nodularis (PN) patients only: Study Design: Subjects meeting study criteria will undergo a 4-week washout period of other therapies that could impact pruritus through the end of the study (including antihistamines, topical steroids, systemic antipruritic therapies or immunosuppressants).
  Interventions: Drug: Abrocitinib
- Chronic Pruritus of Unknown Origin (Experimental): Chronic Pruritus of Unknown Origin (CPUO) patients only: Study Design: Subjects meeting study criteria will undergo a 4-week washout period of other therapies that could impact pruritus through the end of the study (including antihistamines, topical steroids, systemic antipruritic therapies or immunosuppressants).
  Interventions: Drug: Abrocitinib

INTERVENTIONS:
Drug: Abrocitinib — During the study period, subjects will take one Abrocitinib 200 mg tablet once daily orally. Subjects will be directed to take doses of Abrocitinib at approximately the same time of day.

SUMMARY:
The primary objective is to assess the efficacy, safety, and tolerability of Abrocitinib for the treatment of Prurigo Nodularis (PN) or Chronic Pruritus of Unknown Origin (CPUO) in patients experiencing moderate to severe pruritus.

DETAILED DESCRIPTION:
This is a trial to assess the efficacy of Abrocitinib as a therapeutic for Prurigo Nodularis (PN) and Chronic Pruritus of Unknown Origin (CPUO). The study will consist of a 4-week Screening period, a 12-week treatment period and then a 4-week follow up period. The arms will run in parallel and patients will take 200 mg oral Abrocitinib daily for the duration of the 12-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Males or female participants between ages 18-80 years at time of signing informed consent
* A clinical diagnosis of prurigo nodularis, defined by the presence of at least 10 pruritic nodules on at least 2 different anatomic locations (with each arm, leg, and anterior and posterior trunk considered distinct anatomic locations)

OR

* Subject has ongoing chronic pruritus of unknown origin, which must be present on multiple segments on the body. CPUO patients must not have known dermatologic or systemic conditions, that in the opinion of the investigator, are the cause of patient's pruritus
* Subject has moderate to severe pruritus, defined as average peak pruritus numeric rating scale - (PP-NRS) > 7 (range 0-10, higher score indicating greater degree of pruritus severity) in the 7 days prior to the Screening Visit.
* Female participants are eligible for the study if they are not pregnant, planning to become pregnant or breastfeeding during the study or not a woman of child bearing potential (WOCBP)

Exclusion Criteria:

* Infected with hepatitis B or hepatitis C viruses.
* Infected with Herpes Simplex or Herpes zoster.
* Positive HIV serology at screening,
* Evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB)
* History of lymphoproliferative disease, or active primary or recurrent malignancy
* History of recurrent (≥ 2) venous thromboembolism (VTE) or (DVT/PE) - deep vein thrombosis and pulmonary embolism
* Untreated thyroid, adrenal, or pituitary disease or nodules, or history of thyroid malignancy
* Have received any of the following treatment regiments specified in the timeframes outlined below:

  * Within 6 months of first dose of study drug: Rituximab, any other B cell depleting therapies, or intravenous immunoglobulin (IVIg)
  * Within 12 weeks of first dose of study drug: Any studies with Janus kinase (JAK) inhibitors; Cyclophosphamide (or any other cytotoxic agent), belimumab, or anifrolumab (or another anti-interferon (IFN) therapy)
  * Within 8 weeks of first dose of study drug: Other biologics
  * Within 6 weeks: Have been vaccinated with live or attenuated live vaccine.
  * Within 4 weeks: Participation in other studies involving investigational drug(s)
  * Within 4 weeks: Use of oral immune suppressants; systemic immunosuppressive therapies, neuromodulatory therapies, Phototherapy (NB UVB) or broad band phototherapy; Regular use (more than 2 visits per week) of a tanning booth/parlor.
  * Within 1 week of first dose of study drug: Topical treatments that could affect PN; Herbal medications with unknown properties or known beneficial effects for PN.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shawn G Kwatra, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Outpatient Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kwatra SG, Bordeaux ZA, Parthasarathy V, Kollhoff AL, Alajmi A, Pritchard T, Cornman HL, Kambala A, Lee KK, Manjunath J, Ma EZ, Dillen C, Kwatra MM. Efficacy and Safety of Abrocitinib in Prurigo Nodularis and Chronic Pruritus of Unknown Origin: A Nonrandomized Controlled Trial. JAMA Dermatol. 2024 Jul 1;160(7):717-724. doi: 10.1001/jamadermatol.2024.1464. PMID 38837144

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited by referral or at Johns Hopkins Dermatology clinic between September 2021 and March 2022
Pre-assignment Details: 25 patients were assessed for eligibility and screening; four patients failed screening due to laboratory values or presence of uncontrolled disease. One patient left the study voluntarily. Therefore, 20 patients were enrolled in the study
Period: Overall Study
Arm/Group | Prurigo Nodularis | Chronic Pruritus of Unknown Origin
Started | 10 | 10
End of Intervention Period. Week 12: Per Protocol Population | 10 | 10
Follow-up Period (4 Weeks) | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prurigo Nodularis | Chronic Pruritus of Unknown Origin | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (13.1) | 70.7 (5.6) | 64.7 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 2 | 12
  Male | 0 | 8 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 0 | 5
  White | 5 | 10 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Weekly Average Peak Pruritus Numeric Rating Scale (PP-NRS) From Baseline to Week 12
Description: Percent change in weekly average PP-NRS at Week 12. PP-NRS is a single self-report item on an 11-point scale (0 to10) where 0 is No itch, and 10 is the Worst itch imaginable.
Time Frame: Up to 12 weeks
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Prurigo Nodularis | Chronic Pruritus of Unknown Origin
Number analyzed (Participants) | 10 | 10
percent change | -78.26 [-118.48 to -38.09] | -53.66 [-98.76 to -8.55]
Statistical Analysis 1: Comparison: Prurigo Nodularis; Test type: Superiority; p < 0.001, ANOVA — Threshold of significance at 0.05; Mean Difference (Net) = 78.26, 95% CI 2-sided [38.09 to 118.48], Standard Error of Mean 16.15 — Percent PP-NRS reduction comparing subject's values at Week 0 to values at Week 12
Statistical Analysis 2: Comparison: Chronic Pruritus of Unknown Origin; Test type: Superiority; p = 0.0142, ANOVA — Threshold of significance at 0.05; Mean Difference (Net) = 53.66, 95% CI 2-sided [8.55 to 98.76], Standard Error of Mean 18.12 — Percent PP-NRS reduction comparing subject's values at Week 0 to values at Week 12

2. Secondary Outcome: Number of Subjects Achieving a Reduction in Weekly Average PP-NRS From Baseline to Week 12
Description: Number of subjects achieving at least a 4-point reduction from baseline in weekly average PP-NRS at Week 12. The PP-NRS is a single self-report item on an 11-point scale (0 to10) where 0 is No itch, and 10 is the Worst itch imaginable.
Time Frame: Up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prurigo Nodularis | Chronic Pruritus of Unknown Origin
Number analyzed (Participants) | 10 | 10
Participants | 8 | 6

3. Secondary Outcome: Itch Severity Assessed by 5-D Pruritus Scale at Baseline and Week 12
Description: Assess itch severity as assessed by 5-D pruritus scale. The 5-D pruritus scale scores pruritus over the past 2 weeks along 5 dimensions: duration, degree, direction, disability and distribution. Duration, degree and direction are scored from 1 to 5, with "1" indicating better control and resolution of symptoms, and "5" indicating increased intensity, severity and worsening. Disability is assessed in Leisure/Social, housework/errands, and work/school with scores ranging from N/A, and 1-5, with "1" indicating that itch never affects the activity, and "5" meaning that itch always affects this activity. The scores of each of the 5 domains are achieved separately and then summed together to obtain a total score. Scores can range between 5 no pruritus, and 25 most severe pruritus.
Time Frame: Baseline (week 0) and 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Prurigo Nodularis | Chronic Pruritus of Unknown Origin
Number analyzed (Participants) | 10 | 10
score on a scale
  Week 0 | 18.60 [14.98 to 22.22] | 17.40 [14.89 to 19.91]
  Week 12 | 9.20 [7.59 to 10.81] | 11.30 [6.40 to 16.20]
Statistical Analysis 1: Comparison: Prurigo Nodularis; We are comparing baseline scores at Week 0 to scores taken at the end of the treatment period in Week 12; Test type: Superiority; p = 0.002, Wilcoxon matched pairs signed rank test — Threshold of significance at 0.05; Mean Difference (Net) = 9.40, 95% CI 2-sided [6.3 to 12.5], Standard Error of Mean 1.37
Statistical Analysis 2: Comparison: Chronic Pruritus of Unknown Origin; We are comparing baseline scores at Week 0 to scores taken at the end of the treatment period in Week 12; Test type: Superiority; p = 0.0215, Wilcoxon matched pairs signed rank test — Threshold of significance at 0.05; Mean Difference (Net) = 6.10, 95% CI 2-sided [1.6 to 10.6], Standard Error of Mean 1.99

4. Secondary Outcome: Quality of Life as Assessed by the Dermatology Quality of Life Index From Baseline and Week 12
Description: Quality of life as assessed by the Dermatology Quality of Life Index (DLQI). The DLQI is 10 questions used to assess impact of skin disease. Scores range from 0-30, with "0" corresponding to best quality of life, and "30" corresponding to worst quality of life.
Time Frame: Baseline (week 0) and 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Prurigo Nodularis | Chronic Pruritus of Unknown Origin
Number analyzed (Participants) | 10 | 10
score on a scale
  Week 0 | 19.0 [13.30 to 24.70] | 9.60 [6.40 to 12.80]
  Week 12 | 8.90 [4.31 to 13.49] | 4.90 [2.68 to 7.12]
Statistical Analysis 1: Comparison: Prurigo Nodularis; We are comparing baseline scores at Week 0 to scores taken at the end of the treatment period in Week 12; Test type: Superiority; p = 0.002, Wilcoxon matched pairs signed rank test — Threshold of significance at 0.05; Mean Difference (Net) = 10.1, 95% CI 2-sided [5.9 to 14.3], Standard Error of Mean 1.86
Statistical Analysis 2: Comparison: Chronic Pruritus of Unknown Origin; We are comparing baseline scores at Week 0 to scores taken at the end of the treatment period in Week 12; Test type: Superiority; p = 0.02, Wilcoxon matched pairs signed rank test — Threshold of significance at 0.05; Mean Difference (Net) = 4.7, 95% CI 2-sided [0.77 to 8.6], Standard Error of Mean 1.74

5. Secondary Outcome: Pruriginous Lesions as Assessed by the Prurigo Activity Score From Baseline and Week 12
Description: Pruriginous lesions as assessed by the Prurigo Activity Score (PAS). The PAS is a 7-item questionnaire that assesses the number, distribution and activity of pruriginous lesions. The score is calculated via summation of the scoring values, added up with 123 and afterwards divided by 10. This results in a range of values from 1.3 to 21.3.
Time Frame: Baseline (week 0) and 12 weeks
Population: Since this is an assessment for Prurigo Nodularis, only Prurigo Nodularis patients were assessed for this outcome. Data was not collected for patient with Chronic Pruritus of Unknown Origin
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Prurigo Nodularis
Number analyzed (Participants) | 10
score on a scale
  Week 0 | 14.76 [13.04 to 16.48]
  Week 12 | 9.32 [6.57 to 12.07]
Statistical Analysis 1: Comparison: Prurigo Nodularis; We are comparing baseline scores at Week 0 to scores taken at the end of the treatment period in Week 12; Test type: Superiority; p = 0.0078, Wilcoxon matched pairs signed rank test — Threshold of significance at 0.05; Mean Difference (Net) = 5.44, 95% CI 2-sided [2.70 to 8.18], Standard Error of Mean 1.21

6. Secondary Outcome: Itch-scratching Behavior as Assessed by Patient Reported Outcomes Measurement Information System at Baseline and Week 12
Description: Itch-scratching behavior as assessed by Patient Reported Outcomes Measurement Information System (PROMIS®) Itch Questionnaire (PIQ) T-Score: Scratching. The PIQ T-Score: Scratching, is comprised of 5 questions to assess Itch-Scratching Behavior over the past 7 days. Scores for each question range from 1-5, Score range of 5-25 with scores of "1" indicating less scratching behavior and scores of "5" indicating the greatest scratching behavior.
  A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like Itch, a T-score of 60 is one SD worse than average. By comparison, an Itch T-score of 40 is one SD better than average
  For PROMIS, the T-scores have a mean (SD) of 50 (10) for adults in the US experiencing itch for any reason.
Time Frame: Baseline (week 0) and 12 weeks
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Prurigo Nodularis | Chronic Pruritus of Unknown Origin
Number analyzed (Participants) | 10 | 10
T-score
  Week 0 | 53.76 [48.74 to 58.78] | 45.60 [41.57 to 49.63]
  Week 12 | 41.03 [32.67 to 49.39] | 35.72 [30.28 to 41.16]
Statistical Analysis 1: Comparison: Prurigo Nodularis; We are comparing baseline scores at Week 0 to scores taken at the end of the treatment period in Week 12; Test type: Superiority; p = 0.0098, Wilcoxon matched pairs signed rank test — Threshold of significance at 0.05; Mean Difference (Net) = 12.73, 95% CI 2-sided [5.57 to 19.89], Standard Error of Mean 3.16
Statistical Analysis 2: Comparison: Chronic Pruritus of Unknown Origin; We are comparing baseline scores at Week 0 to scores taken at the end of the treatment period in Week 12; Test type: Superiority; p = 0.0117, Wilcoxon matched pairs signed rank test — Threshold of significance at 0.05; Mean Difference (Net) = 9.88, 95% CI 2-sided [3.10 to 16.66], Standard Error of Mean 3.00

7. Secondary Outcome: Number of Nodules at Baseline and Week 12
Description: Number of baseline prurigo nodules over time. As part of the Prurigo Activity Score, lesions are counted in a representative body region. Lesion count within the representative area at Week 0 was compared to lesion count in the representative area at Week 12.
Time Frame: Baseline (week 0) and 12 weeks
Population: Assessed only in participants with nodules (Prurigo Nodularis arm). Since this is an assessment for Prurigo Nodularis, only Prurigo Nodularis patients were assessed for this outcome. Data was not collected for patient with Chronic Pruritus of Unknown Origin.
Measure: Mean (95% Confidence Interval); unit: Lesion count
Arm/Group | Prurigo Nodularis
Number analyzed (Participants) | 10
Lesion count
  Week 0 | 14.90 [9.21 to 20.59]
  Week 12 | 4.70 [2.59 to 6.81]
Statistical Analysis 1: Comparison: Prurigo Nodularis; We are comparing baseline scores at Week 0 to scores taken at the end of the treatment period in Week 12; Test type: Superiority; p = 0.002, Wilcoxon matched pairs signed rank test — Threshold of significance at 0.05; Mean Difference (Net) = 10.20, 95% CI 2-sided [4.46 to 15.94], Standard Error of Mean 2.54

8. Secondary Outcome: Prurigo Nodule Severity at Baseline and Week 12
Description: Prurigo nodule severity using the Investigator's Global Assessment (IGA). The IGA is a physician scale assessing the number of nodules a Prurigo Nodularis (PN) patient has. Patients receive a score between 0 and 4, where "0" is clear: "No prurigo nodules. Post-inflammatory hypo/hyper pigmentation may be present". Grades of "4" are severe: "Abundant prurigo nodules. Marked nodule elevation."
Time Frame: Baseline (week 0) and 12 weeks
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Prurigo Nodularis
Number analyzed (Participants) | 10
score on a scale
  Week 0 | 3.60 [3.23 to 3.97]
  Week 12 | 2.50 [1.99 to 3.01]
Statistical Analysis 1: Comparison: Prurigo Nodularis; We are comparing baseline scores at Week 0 to scores taken at the end of the treatment period in Week 12; Test type: Superiority; p = 0.0078, Wilcoxon matched pairs signed rank test — Threshold of significance at 0.05; Mean Difference (Net) = 1.10, 95% CI 2-sided [0.57 to 1.63], Standard Error of Mean 0.23

9. Secondary Outcome: Quality of Life as Assessed by the EuroQoL 5-Dimension at Baseline and Week 12
Description: Quality of life as assessed by EuroQoL 5-Dimension (EQ-5D). The 3 level version of the EQ-5D (EQ-5D-3L) assesses degree of debilitation in 5 major aspects of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has three possible answers. These answers equate to: "No problems" or "Some/Moderate Problems" or "Severe/Extreme problems. The patient is asked to indicate their health state by ticking the box next to the most appropriate statement in each of the five dimensions. A unique health state is then defined by combining one level from each of the 5 dimensions. Each state is referred to in terms of a 5-digit code. A total of 243 possible health states codes is defined in this way. State 11111 indicates no problems on any of the five dimensions. The patient then rates how good or bad their health is on that day from a range from 0 the worst health you can imagine, to 100 the best health you can imagine.
Time Frame: Baseline (week 0) and 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Prurigo Nodularis | Chronic Pruritus of Unknown Origin
Number analyzed (Participants) | 10 | 10
score on a scale
  Week 0 | 0.60 [0.33 to 0.87] | 0.74 [0.55 to 0.93]
  Week 12 | 0.75 [0.52 to 0.99] | 0.86 [0.67 to 1.05]
Statistical Analysis 1: Comparison: Prurigo Nodularis; We are comparing baseline scores at Week 0 to scores taken at the end of the treatment period in Week 12; Test type: Superiority; p = 0.0391, Wilcoxon matched pairs signed rank test — Threshold of significance at 0.05; Mean Difference (Net) = 0.15, 95% CI 2-sided [0.025 to 0.27], Standard Error of Mean 0.055
Statistical Analysis 2: Comparison: Chronic Pruritus of Unknown Origin; We are comparing baseline scores at Week 0 to scores taken at the end of the treatment period in Week 12; Test type: Superiority; p = 0.28, Wilcoxon matched pairs signed rank test — Threshold of significance at 0.05; Mean Difference (Net) = 0.12, 95% CI 2-sided [-.080 to 0.31], Standard Error of Mean 0.086

10. Secondary Outcome: Depression as Assessed by The Hospital Anxiety and Depression Scale at Baseline and Week 12
Description: Depression as assessed by The Hospital Anxiety and Depression Scale (HADS), has 7 items relating to depression. Each item scored from 0-3 with higher scores indicating higher depression. Total score range 0-21.
Time Frame: Baseline (week 0) and 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Prurigo Nodularis | Chronic Pruritus of Unknown Origin
Number analyzed (Participants) | 10 | 10
score on a scale
  Week 0 | 6.90 [3.42 to 10.38] | 4.20 [0.93 to 7.47]
  Week 12 | 3.30 [0.398 to 6.202] | 3.10 [0.310 to 5.890]
Statistical Analysis 1: Comparison: Prurigo Nodularis; We are comparing baseline scores at Week 0 to scores taken at the end of the treatment period in Week 12; Test type: Superiority; p = 0.0684, Wilcoxon matched pairs signed rank test — Threshold of significance at 0.05; Mean Difference (Net) = 3.6, 95% CI 2-sided [0.035 to 7.235], Standard Error of Mean 1.607
Statistical Analysis 2: Comparison: Chronic Pruritus of Unknown Origin; Test type: Superiority; p = 0.375, Wilcoxon matched pairs signed rank test — Threshold of significance at 0.05; Mean Difference (Net) = 1.10, 95% CI 2-sided [-3.656 to 1.456], Standard Error of Mean 1.13

11. Secondary Outcome: Anxiety as Assessed by The Hospital Anxiety and Depression Scale at Baseline and Week 12
Description: Anxiety as assessed by The Hospital Anxiety and Depression Scale (HADS), has 7 items relating to anxiety. Each item scored from 0-3 with higher scores indicating higher anxiety. Total score range 0-21.
Time Frame: Baseline (week 0) and 12 weeks
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Prurigo Nodularis | Chronic Pruritus of Unknown Origin
Number analyzed (Participants) | 10 | 10
score on a scale
  Week 0 | 6.60 [2.62 to 10.58] | 4.30 [0.061 to 8.54]
  Week 12 | 5.90 [2.61 to 9.20] | 4.30 [0.27 to 8.33]
Statistical Analysis 1: Comparison: Prurigo Nodularis; We are comparing baseline scores at Week 0 to scores taken at the end of the treatment period in Week 12; Test type: Superiority; p = 0.207, Wilcoxon matched pairs signed rank test — Threshold of significance at 0.05; Mean Difference (Net) = 0.70, 95% CI 2-sided [-3.44 to 2.04], Standard Error of Mean 1.212
Statistical Analysis 2: Comparison: Chronic Pruritus of Unknown Origin; We are comparing baseline scores at Week 0 to scores taken at the end of the treatment period in Week 12; Test type: Superiority; p = 0.8125, Wilcoxon matched pairs signed rank test — Threshold of significance at 0.05; Mean Difference (Net) = 0, 95% CI 2-sided [-3.389 to 3.389], Standard Error of Mean 1.498

12. Secondary Outcome: Sleep Disturbance as Assessed by the SD-NRS at Baseline and Week 12
Description: Average sleep disturbance from Week 0 and Week 12 as assessed by (SD) NRS. The SD-NRS is an 11-point scale (0 -10) with higher scores indicating greater sleep disturbance.
Time Frame: Baseline (week 0) and 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Prurigo Nodularis | Chronic Pruritus of Unknown Origin
Number analyzed (Participants) | 10 | 10
score on a scale
  Week 0 | 7.20 [5.52 to 8.88] | 5.10 [2.66 to 7.54]
  Week 12 | 2.40 [-0.060 to 4.86] | 2.80 [-0.017 to 5.62]
Statistical Analysis 1: Comparison: Prurigo Nodularis; We are comparing baseline scores at Week 0 to scores taken at the end of the treatment period in Week 12; Test type: Superiority; p = 0.0039, Wilcoxon matched pairs signed rank test — Threshold of significance at 0.05; Mean Difference (Net) = 4.80, 95% CI 2-sided [2.52 to 7.08], Standard Error of Mean 1.009
Statistical Analysis 2: Comparison: Chronic Pruritus of Unknown Origin; We are comparing baseline scores at Week 0 to scores taken at the end of the treatment period in Week 12; Test type: Superiority; p = 0.0547, Wilcoxon matched pairs signed rank test — Threshold of significance at 0.05; Mean Difference (Net) = 2.3, 95% CI 2-sided [-0.0376 to 4.638], Standard Error of Mean 1.033

13. Secondary Outcome: Itch Intensity in Patients With Underlying Atopy at Baseline and Week 12
Description: Itch intensity as assessed by PP-NRS in Prurigo Nodularis patients with underlying atopy. The PP-NRS is a single self-report item on an 11-point scale (0 to10) where 0 is No itch, and 10 is the Worst itch imaginable. Atopy defined as a binary variable where patients have 2 out of 3: underlying history of atopic dermatitis, history of seasonal allergies, or asthma.
Time Frame: Baseline (week 0) and 12 weeks
Population: Prurigo Nodularis patients with underlying atopy
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Prurigo Nodularis
Number analyzed (Participants) | 3
score on a scale
  Week 0 | 9.67 [8.23 to 11.10]
  Week 12 | 0.67 [-2.20 to 3.54]
Statistical Analysis 1: Comparison: Prurigo Nodularis; We are comparing baseline scores at Week 0 to scores taken at the end of the treatment period in Week 12; Test type: Superiority; p = 0.0003, t-test, 2 sided — Threshold of significance at 0.05; Mean Difference (Net) = 9.00, 95% CI 2-sided [6.93 to 11.07]

14. Secondary Outcome: Itch Intensity in Patients Without Underlying Atopy at Baseline and Week 12
Description: Itch intensity as assessed by PP-NRS in Prurigo Nodularis patients without underlying atopy. The PP-NRS is a single self-report item on an 11-point scale (0 to10) where 0 is No itch, and 10 is the Worst itch imaginable. Atopy is defined as a binary variable where patients have 2 out of 3: underlying history of atopic dermatitis, history of seasonal allergies, or asthma.
Time Frame: Baseline (week 0) and 12 weeks
Population: Prurigo Nodularis patients without underlying atopy
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Prurigo Nodularis
Number analyzed (Participants) | 7
score on a scale
  Week 0 | 9.00 [7.93 to 10.07]
  Week 12 | 2.57 [0.075 to 5.07]
Statistical Analysis 1: Comparison: Prurigo Nodularis; Test type: Superiority; p < 0.0001, t-test, 2 sided — Threshold of significance at 0.05; Mean Difference (Net) = 6.429, 95% CI 2-sided [4.011 to 8.846]

15. Secondary Outcome: Itch Intensity in CPUO Patients With High Eosinophilia at Baseline and Week 12
Description: Itch intensity as measured by PP-NRS in CPUO patients with high eosinophilia (greater than 500 eosinophils per micro-liter of blood). The PP-NRS is an 11-point single self-report item on a scale (0 to10) where 0 is No itch, and 10 is the Worst itch imaginable.
Time Frame: Baseline (week 0) and 12 weeks
Population: Data not collected. None of the CPUO subjects met the pre-defined criteria for eosinophilia.
Arm/Group | Chronic Pruritus of Unknown Origin
Number analyzed (Participants) | 0

16. Secondary Outcome: Cutaneous Biomarker Analysis - Gene Set Variation Analysis (GSVA), at Baseline and Week 12
Description: Lesional and non-lesional skin biopsies will be compared for Type 1/2/17/22 T Helper (Th) Th1/Th2/Th17/Th22 polarization before and after treatment. PN and CPUO patients had biopsies collected at Week 0 and at Week 12. PN patients had two biopsies collected: a lesional site and a non-lesional biopsy close by for comparison. The CPUO patients only had one biopsy collected at the timepoints because there are no visible lesions.
  CPUO will be compared from week 0 to week 12. PN will compare Lesional to non Lesional at Week 0. PN will compare Lesional to Non Lesional at Week 12.
  GSVA will compare gene set enrichment scores as a function of gene pathway expression which range from -1 to 1. Lower scores indicate down regulation of the gene set, and higher scores indicate up regulation.
Time Frame: Baseline (week 0) and 12 weeks
Population: PN and CPUO patients had biopsies collected at Week 0 and at Week 12. PN patients had two biopsies collected: a lesional site and a non-lesional biopsy close by for comparison. The CPUO patients only had one biopsy collected at the timepoints because there are no visible lesions.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Prurigo Nodularis | Chronic Pruritus of Unknown Origin
Number analyzed (Participants) | 10 | 10
score on a scale
  Th1 Lesional Week 0 | 0.35 [0.0035 to 0.69] | 0.27 [0.076 to 0.46]
  Th1 Non Lesional Week 0: number analyzed (Participants) | 10 | 0
  Th1 Non Lesional Week 0 | -0.085 [-0.31 to 0.14] |
  Th1 Lesional Week 12 | 0.045 [-0.31 to 0.40] | -0.31 [-0.49 to -0.14]
  Th1 Non Lesional Week 12: number analyzed (Participants) | 10 | 0
  Th1 Non Lesional Week 12 | -0.36 [-0.70 to -0.021] |
  Th2 Lesional Week 0 | 0.22 [-0.047 to 0.49] | 0.17 [0.016 to 0.32]
  Th2 Non Lesional Week 0: number analyzed (Participants) | 10 | 0
  Th2 Non Lesional Week 0 | -0.11 [-0.31 to 0.086] |
  Th2 Lesional Week 12 | 0.10 [-0.16 to 0.37] | -0.20 [-0.32 to -0.083]
  Th2 Non Lesional Week 12: number analyzed (Participants) | 10 | 0
  Th2 Non Lesional Week 12 | -0.18 [-0.44 to 0.080] |
  Th17 Lesional Week 0 | 0.29 [0.048 to 0.52] | 0.12 [-0.10 to 0.33]
  Th17 Non Lesional Week 0: number analyzed (Participants) | 10 | 0
  Th17 Non Lesional Week 0 | -0.29 [-0.52 to -0.062] |
  Th17 Lesional Week 12 | 0.20 [-0.16 to 0.57] | -0.099 [-0.25 to 0.050]
  Th17 Non Lesional Week 12: number analyzed (Participants) | 10 | 0
  Th17 Non Lesional Week 12 | -0.083 [-0.45 to 0.29] |
  Th22 Lesional Week 0 | 0.23 [-0.060 to 0.52] | 0.23 [0.048 to 0.42]
  Th22 Non Lesional Week 0: number analyzed (Participants) | 10 | 0
  Th22 Non Lesional Week 0 | -0.29 [-0.50 to -0.071] |
  Th22 Lesional Week 12 | 0.25 [-0.060 to 0.55] | -0.15 [-0.34 to 0.034]
  Th22 Non Lesional Week 12: number analyzed (Participants) | 10 | 0
  Th22 Non Lesional Week 12 | -0.16 [-0.49 to 0.17] |
Statistical Analysis 1: Comparison: Chronic Pruritus of Unknown Origin; This is a comparison of Th1 GSVA from RNA sequencing (RNASeq) performed on skin biopsies. The comparison is for CPUO patient skin at Week 0 versus Week 12 (end of treatment) The CPUO patients only had one biopsy collected at the timepoints because there are no visible lesions. CPUO patients only had one biopsy taken which will be referred to as Lesional sites. CPUO will compare Lesional biopsies at week 0 to Lesional biopsies at week 12; Test type: Superiority; p < 0.0001, t-test, 2 sided — Threshold of significance set at 0.05; Median Difference (Net) = -0.58, 95% CI 2-sided [-0.83 to -0.33], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Chronic Pruritus of Unknown Origin; This is a comparison of Th2 GSVA from RNASeq performed on skin biopsies. The comparison is for CPUO patient skin at Week 0 versus Week 12 (end of treatment) The CPUO patients only had one biopsy collected at the timepoints because there are no visible lesions. CPUO patients only had one biopsy taken which will be referred to as Lesional sites. CPUO will compare Lesional biopsies at week 0 to Lesional biopsies at week 12; Test type: Superiority; p = 0.0003, t-test, 2 sided — The threshold for significance is set at 0.05; Mean Difference (Net) = -0.37, 95% CI 2-sided [-0.56 to -0.18], Standard Error of Mean 0.091
Statistical Analysis 3: Comparison: Chronic Pruritus of Unknown Origin; This is a comparison of Th17 GSVA from RNASeq performed on skin biopsies. The comparison is for CPUO patient skin at Week 0 versus Week 12 (end of treatment) The CPUO patients only had one biopsy collected at the timepoints because there are no visible lesions. CPUO patients only had one biopsy taken which will be referred to as Lesional sites. CPUO will compare Lesional biopsies at week 0 to Lesional biopsies at week 12; Test type: Superiority; p = 0.0952, t-test, 2 sided — The threshold for significance is set at 0.05; Mean Difference (Net) = -0.21, 95% CI 2-sided [-0.47 to 0.039], Standard Error of Mean 0.12
Statistical Analysis 4: Comparison: Chronic Pruritus of Unknown Origin; This is a comparison of Th22 GSVA from RNASeq performed on skin biopsies. The comparison is for CPUO patient skin at Week 0 versus Week 12 (end of treatment) The CPUO patients only had one biopsy collected at the timepoints because there are no visible lesions. CPUO patients only had one biopsy taken which will be referred to as Lesional sites. CPUO will compare Lesional biopsies at week 0 to Lesional biopsies at week 12; Test type: Superiority; p = 0.004, t-test, 2 sided — Threshold for significance is set at 0.05; Mean Difference (Net) = -0.38, 95% CI 2-sided [-0.64 to -0.13], Standard Error of Mean 0.12
Statistical Analysis 5: Comparison: Prurigo Nodularis; This is a comparison of Th1 GSVA from RNASeq performed on skin biopsies. The comparison is for lesional PN patient skin at Week 0 versus non lesional PN patient skin at week 0; Test type: Superiority; p = 0.0277, t-test, 2 sided — The threshold of significance is set at 0.05; Mean Difference (Net) = -0.43, 95% CI 2-sided [-0.81 to -0.053], Standard Error of Mean 0.18
Statistical Analysis 6: Comparison: Prurigo Nodularis; This is a comparison of Th1 GSVA from RNASeq performed on skin biopsies. The comparison is for lesional PN patient skin at Week 12 versus non lesional PN patient skin at week 12; Test type: Superiority; p = 0.077, t-test, 2 sided — The threshold of significance is set at 0.05; Mean Difference (Net) = -0.40, 95% CI 2-sided [-0.85 to 0.049], Standard Error of Mean 0.22
Statistical Analysis 7: Comparison: Prurigo Nodularis; This is a comparison of Th2 GSVA from RNASeq performed on skin biopsies. The comparison is for lesional PN patient skin at Week 0 versus non lesional PN patient skin at Week 0; Test type: Superiority; p = 0.0363, t-test, 2 sided — The threshold of significance is set at 0.05; Mean Difference (Net) = -0.33, 95% CI 2-sided [-0.64 to -0.024], Standard Error of Mean 0.15
Statistical Analysis 8: Comparison: Prurigo Nodularis; This is a comparison of Th2 GSVA from RNASeq performed on skin biopsies. The comparison is for lesional PN patient skin at Week 12 versus non lesional PN patient skin at Week 12; Test type: Superiority; p = 0.10, t-test, 2 sided — The threshold of significance is set at 0.05; Mean Difference (Net) = -0.29, 95% CI 2-sided [-0.63 to 0.062], Standard Error of Mean 0.17
Statistical Analysis 9: Comparison: Prurigo Nodularis; This is a comparison of Th17 GSVA from RNASeq performed on skin biopsies. The comparison is for lesional PN patient skin at Week 0 versus non lesional PN patient skin at Week 0; Test type: Superiority; p = 0.0009, t-test, 2 sided — The threshold for significance is set at 0.05; Mean Difference (Net) = -0.58, 95% CI 2-sided [-0.89 to -0.27], Standard Error of Mean 0.15
Statistical Analysis 10: Comparison: Prurigo Nodularis; This is a comparison of Th17 GSVA from RNASeq performed on skin biopsies. The comparison is for lesional PN patient skin at Week 12 versus non lesional PN patient skin at Week 12; Test type: Superiority; p = 0.2326, t-test, 2 sided — The threshold for significance is set at 0.05; Mean Difference (Net) = -0.28, 95% CI 2-sided [-0.77 to 0.20], Standard Error of Mean 0.23
Statistical Analysis 11: Comparison: Prurigo Nodularis; This is a comparison of Th22 GSVA from RNASeq performed on skin biopsies. The comparison is for lesional PN patient skin at Week 0 versus non lesional PN patient skin at Week 0; Test type: Superiority; p = 0.0047, t-test, 2 sided — The threshold for significance is set at 0.05; Mean Difference (Net) = -0.52, 95% CI 2-sided [-0.85 to -0.18], Standard Error of Mean 0.16
Statistical Analysis 12: Comparison: Prurigo Nodularis; This is a comparison of Th22 GSVA from RNASeq performed on skin biopsies. The comparison is for lesional PN patient skin at Week 12 versus non lesional PN patient skin at Week 12; Test type: Superiority; p = 0.0539, t-test, 2 sided — The threshold for significance is set at 0.05; Mean Difference (Net) = -0.41, 95% CI 2-sided [-0.83 to 0.0076], Standard Error of Mean 0.20

17. Secondary Outcome: Systemic Biomarker Analysis - Gene Set Variation Analysis (GSVA), at Baseline and Week 12
Description: Plasma cytokines will be analyzed for TH1/Th2/Th17/Th22 polarization before and after treatment. This outcome was posted in error. It is not appropriate to perform GSVA of plasma cytokines. It is best practice to limit GSVA to RNASeq.
Time Frame: Baseline and 12 weeks
Population: This outcome was not assessed. Data was not collected.
Arm/Group | Prurigo Nodularis | Chronic Pruritus of Unknown Origin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first date of abrocitinib administration to the last date of abrocitinib administration + 4 week follow up, up to 16 weeks total.
Arm/Group | Prurigo Nodularis | Chronic Pruritus of Unknown Origin
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prurigo Nodularis (N=10) | Chronic Pruritus of Unknown Origin (N=10)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Folliculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Acneiform Eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Sore throat (Infections and infestations) | 1 (1) | 0 (0)
Herpes Labialis (Infections and infestations) | 0 (0) | 1 (1)
Nasal Congestion (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/82/NCT05038982/Prot_SAP_002.pdf
  • Informed Consent Form (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/82/NCT05038982/ICF_003.pdf